CLINICAL TRIAL: NCT01382797
Title: A Phase 2b Randomized, Double-blind, Placebo-controlled, Repeat-dose Study to Evaluate the Safety, Tolerability, and Efficacy of ALKS 37 in Subjects With Opioid-induced Constipation
Brief Title: ALK37-005: A Study of ALKS 37 (RDC-1036) in Adults With Opioid-induced Constipation (OIC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK37-005
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Opioid-induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Capsules for oral administration
  Interventions: Drug: Placebo
- ALKS 37 (Experimental): Capsules for oral administration
  Interventions: Drug: ALKS 37

INTERVENTIONS:
Drug: ALKS 37 — Capsules for oral administration
  Arms: ALKS 37
Drug: Placebo — Capsules for oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of ALKS 37 when administered daily for 4 weeks to adults with Opioid-induced Constipation (OIC).

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age at time of consent
* Have a body mass index (BMI)of 19 to 35 kg/m2 at screening
* Are receiving prescribed opioid medication for the management of chronic, non-cancer pain
* Meet the criteria of OIC
* Agree to use an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* Pregnancy and/or currently breastfeeding
* Clinically significant medical condition or illness (other than the condition for which the pain medication is being prescribed)
* Receiving treatment with opioid therapy for cancer-related pain, abdominal pain, scleroderma, and/or for the management of drug addiction
* Any gastrointestinal (GI) disorder (other than opioid-induced constipation) or GI structural abnormality known to affect bowel transit, produce GI obstruction, or contribute to bowel dysfunction
* Use of naloxone, Subutex or Suboxone, Revia, Relistor, or Entereg starting 15 days before the first study visit following screening until the end of the study
* Participation in a clinical trial of a pharmacological agent within 30 days before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Dose response relationship among five doses of study drug (4 doses of ALKS 37 and placebo), defined as an increasing proportion of patients exhibiting overall response. | 4 weeks
  Overall response will be defined using an algorithm that takes into consideration number of complete spontaneous bowel movements, improvement from baseline, and durability of response.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leigh-Pemberton, M.D., Study Director — Alkermes, Inc.
Locations (20):
- United States (20):
  - Alkermes Study Site, Mesa, Arizona
  - Alkermes Study Site, Phoenix, Arizona
  - Alkermes Study Site, National City, California
  - Alkermes Study Site, Oceanside, California
  - Alkermes Study Site, Pasadena, California
  - Alkermes Study Site, Denver, Colorado
  - Alkermes Investigational Site, DeLand, Florida
  - Alkermes Study Site, Ormond Beach, Florida
  - Alkermes Study Site, St. Petersburg, Florida
  - Alkermes Study Site, Stockbridge, Georgia
  - Alkermes Study Site, Boise, Idaho
  - Alkermes Study Site, New Orleans, Louisiana
  - Alkermes Study Site, Kalamazoo, Michigan
  - Alkermes Study Site, Las Vegas, Nevada
  - Alkermes Study Site, Belvidere, New Jersey
  - Alkermes Study Site, Brooklyn, New York
  - Alkermes Study Site, Cincinnati, Ohio
  - Alkermes Study Site, Oklahoma City, Oklahoma
  - Alkermes Study Site, Medford, Oregon
  - Alkermes Study Site, San Antonio, Texas